CLINICAL TRIAL: NCT00532090
Title: Multiple Ascending Dose (MAD) Study of R4733 Administered Orally in Patients With Refractory Metastatic or Locally Advanced Solid Tumors
Brief Title: A Multiple Ascending Dose Study of R4733 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO21321
Record Dates: First submitted 2007-09-18; First posted 2007-09-19 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RG4733
- 2 (Experimental)
  Interventions: Drug: RG4733
- 3 (Experimental)
  Interventions: Drug: RG4733

INTERVENTIONS:
Drug: RG4733 — Administered orally daily at ascending doses to successive cohorts of patients
  Other Names: RO4929097
  Arms: 3
Drug: RG4733 — Administered orally at ascending doses to successive cohorts of patients, on a 3 days on/ 4 days off schedule
  Other Names: RO4929097
  Arms: 1
Drug: RG4733 — Administered orally at ascending doses to successive cohorts of patients, on days 1-7 of each 21 day cycle
  Other Names: RO4929097
  Arms: 2

SUMMARY:
This study will determine the maximum tolerated dose, safety and pharmacokinetic profile of R4733 (RO4929097), administered orally to patients with refractory metastatic or locally advanced solid tumors. The study will assess three different dosing schedules; in one schedule R4733 will be administered 3days on/ 4 days off, in another on days 1-7 of each 21 day cycle, and in a third schedule continuously daily. The starting dose for each dosing regimen will be escalated in subsequent groups of patients after a satisfactory assessment of the safety and tolerability of the previous dose. The anticipated time on study treatment is until disease progression or dose-limiting toxicity, and the target sample size is 100-200 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* advanced and/or metastatic solid tumor malignancy;
* measurable or evaluable disease;
* ECOG performance status 0 or 1.

Exclusion Criteria:

* prior chemotherapy, radiotherapy or immunotherapy within 28 days of first receipt of study drug;
* prior corticosteroids as anti-cancer therapy within a minimum of 14 days of first receipt of study drug. Dexamethasone may be allowed only as part of the supportive care measures;
* major surgery within 28 days of first receipt of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2007-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters. | Throughout study

SECONDARY OUTCOMES:
Tumor assessments | day 15 cycle 1, at the end of cycle 2 and every 6 weeks thereafter
Pharmacokinetic profile | After first dose and last dose (or day 15) of cycles 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- United States (5):
  - Aurora, Colorado
  - Boston, Massachusetts
  - New Brunswick, New Jersey
  - Houston, Texas
  - San Antonio, Texas